CLINICAL TRIAL: NCT02475421
Title: Hyperglucagonaemia in Patients With Type 2 Diabetes - Role of Glucagon Clearance
Acronym: MCR Glucagon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Principal Investigator, Asger Lund, Asger Lund, MD, PhD-student, University Hospital, Gentofte, Copenhagen, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-1-2014-066
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Diabetes
Keywords: Diabetes; Glucagon; Metabolic clearance rate of glucagon
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy, lean subjects (Experimental): Healthy subjects with BMI < 27 kg/m^2
  Interventions: Biological: Glucagon
- Healthy, obese subjects (Experimental): Healthy subjects with BMI > 33 kg/m^2
  Interventions: Biological: Glucagon
- Diabetic, lean subjects (Experimental): Diabetic subjects with BMI < 27 kg/m^2
  Interventions: Biological: Glucagon
- Diabetic, obese subjects (Experimental): Diabetic subjects with BMI > 33 kg/m^2
  Interventions: Biological: Glucagon

INTERVENTIONS:
Biological: Glucagon — One hour glucagon-clamp followed by one hour of blood sampling

SUMMARY:
The study aims to evaluate the elimination and degradation of glucagon in patients with type 2 diabetes compared to matched healthy subjects.

DETAILED DESCRIPTION:
In the present project the investigators wish to identify whether the elimination and degradation of glucagon differ between healthy control subjects and patients with type 2 diabetes. Furthermore, the investigators wish to examine whether obesity is an independent factor for altered glucagon metabolism. Thus, by examining glucagon elimination in obese subjects with and without type 2 diabetes and in lean subjects with and without type 2 diabetes the investigators will be able to describe the metabolic clearance rate (MCR) of glucagon in a broad spectrum of individuals with different levels of insulin resistance and beta cell dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes

* Caucasians above 35 years of age with diet or/and metformin-treated type 2 diabetes of at least 3 month duration (diagnosed according to World Health Organization (WHO) criteria
* BMI either below 27 or above 33 kg/m^2
* Normal haemoglobin
* Informed consent

Subjects with NGT

* Caucasians above 35 years of age
* BMI either below 27 or above 33 kg/m^2
* Normal HbA1c (according to WHO criteria)
* Normal haemoglobin
* Informed consent

Exclusion Criteria:

Patients with type 2 diabetes

* Inflammatory bowel disease
* Operation within the last 3 months
* Severe kidney disease (eGFR < 60 ml/min)
* Severe liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2×normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years
* Any condition that the investigators feel would interfere with trial participation

Subjects with NGT

* Diabetes
* Prediabetes (impaired FPG or HbA1c above 42 mmol/mol)
* First-degree relatives with diabetes
* Inflammatory bowel disease
* Intestinal resection
* Severe kidney disease (eGFR < 60 ml/min)
* Liver disease (ALA T and/or serum ASA T >2×normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years Any condition that the investigators feel would interfere with trial participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Metabolic clearance rate of glucagon | -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes

SECONDARY OUTCOMES:
Gut and pancreatic hormones | -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
Blood glucose | -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
Basic metabolic rate | -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
Satiety, hunger, appetite - measured with visual analogue scales (VAS) | -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
Half life of glucagon | -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes
The volume of distribution of glucagon | -30, -15, 0, 5, 10, 20, 50, 55, 60, 62, 64, 66, 68, 70, 75, 80, 85, 90, 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Department of Medicine, Gentofte Hospital, Hellerup, Copenhagen, Denmark